CLINICAL TRIAL: NCT03485118
Title: Phase II Study on Safety and Efficacy of Recombinant Human-mouse Chimeric Anti-CD20 Monoclonal Antibody (HS006) Combined With CHOP (Hi-CHOP) in Patients With Previously Untreated Diffuse Large B-cell Lymphoma
Brief Title: RHCACD20MA (HS006) Combined With CHOP (Hi-CHOP) in Patients With Previously Untreated Diffuse Large B-cell Lymphoma
Acronym: Hi-CHOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HISUN-CD20-2016L01
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Previously untreated DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, controlled, multicenter phase II study.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS006+Chemotherapy (Experimental): 1. Participants received six 21-day cycles of HS006(375 mg per square meter) combined with six cycles of standard cyclophosphamide,doxorubicin,vincristine,and prednisone/prednisolone(CHOP) chemotherapy(21-day cycles).
  2. Participants received six 21-day cycles of HS006(500 mg per square meter) combined with six cycles of standard cyclophosphamide,doxorubicin,vincristine,and prednisone(CHOP) chemotherapy(21-day cycles).
  Interventions: Drug: HS006+CHOP
- Rituxan+Chemotherapy (Active Comparator): Participants received six 21-day cycles of Rituxan combined with six cycles of standard cyclophosphamide,doxorubicin,vincristine,and prednisone(CHOP) chemotherapy(21-day cycles).
  Interventions: Drug: Rituximab+CHOP

INTERVENTIONS:
Drug: HS006+CHOP — Drug:HS006 HS006 375 mg per square meter (mg/m^2),administered intravenously(IV) on Day1 of each 21-day cycle for 6 cycles.
  Drug :Cyclophosphamide Cyclophosphamide 750mg per square metre(mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Doxorubicin Doxorubicin 50mg per square metre( mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Vincristine Vincristine 1.4mg(maximum 2.0mg) per square metre (mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug: Prednisone Prednisone 100 mg administered orally on Days 2-6 of each 21-day cycle.
  Arms: HS006+Chemotherapy
Drug: HS006+CHOP — Drug:HS006 HS006 500 mg per square meter (mg/m^2),administered intravenously(IV) on Day1 of each 21-day cycle for 6 cycles. During cycle 1,HS006 also infused on Day 8 and 15.
  Drug :Cyclophosphamide Cyclophosphamide 750mg per square metre(mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Doxorubicin Doxorubicin 50mg per square metre( mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Vincristine Vincristine 1.4mg(maximum 2.0mg) per square metre (mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug: Prednisone Prednisone 100 mg administered orally on Days 1-5 of each 21-day cycle.
  Arms: HS006+Chemotherapy
Drug: Rituximab+CHOP — Drug:Rituxan Rituxan 375 mg per square metre (mg/m^2), administered by intravenous (IV) on Day 1 of each 21-day cycle.
  Drug :Cyclophosphamide Cyclophosphamide 750mg per square metre(mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Doxorubicin Doxorubicin 50mg per square metre( mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug :Vincristine Vincristine 1.4mg(maximum 2.0mg) per square metre (mg/m^2),administered intravenously(IV) on Day 2 of each 21-day cycle.
  Drug: Prednisone Prednisone 100 mg administered orally on Days 2-6 of each 21-day cycle.
  Arms: Rituxan+Chemotherapy

SUMMARY:
Primary objective:

To evaluate the efficacy of recombinant human-mouse chimeric anti-CD20 monoclonal antibody injection(HS006) with CHOP(Hi-CHOP) versus Rituximab with CHOP (R-CHOP) in patients with previously untreated Diffuse Large B-cell Lymphoma as first line treatment.

Secondary objective:

To evaluate the safety of recombinant human-mouse chimeric anti-CD20 monoclonal antibody injection(HS006) with CHOP(Hi-CHOP) in patients with previously untreated Diffuse Large B-cell Lymphoma.

To study the pharmacokinetics of recombinant human-mouse chimeric anti-CD20 monoclonal antibody injection(HS006) in patients with previously untreated Diffuse Large B-cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. previously untreated. CD20 Positive DLBCL.
2. Lymphoma International PrognosisIndex (IPI) score of 0-3, stage I-IV.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2, Expected survival>6 months.
4. At least 1 bi-dimensionally measurable lesion: Nodal lesion: Greatest transverse diameter ≥1.5cm and short axis ≥1.0cm; Extra-nodal lesion: Greatest transverse diameter≥1.0cm.
5. CBC: WBC >4 x 10^9/L;NEU > 2 x 10^9 / L; PLT > 100 x 10^9 / L; Patients with bone marrow infiltration: WBC≥3 x 10^9/L、HGB≥80g/L、NEU≥1.5 x 10^9/L、PLT≥75 x 10^9/L；
6. hepatic function: TBIL≤1.5 x ULN；ALT or AST ≤2.5 x ULN； ALP≤3 x ULN if with no bone marrow infiltration;Renal function: Cr≤1.5 x ULN；
7. HIV negative;
8. HCV-Ab negative OR HCV-Ab positive but HCV-RNA negative.
9. HBsAg and HBcAb negative,HBsAg or HBcAb positive with HBV DNA<1×1000IU / ml.
10. Cardiac echocardiography :LVEF ≥ 50%;
11. Must agree to take effective birth control methods or are not of childbearing potential. Women must agree to continue contraceptive measures within 12 months after the last treatment. Men must agree to continue contraception within 3 months after the treatment.
12. All patients must have signed an informed consent document.

Exclusion Criteria:

1. Patients with primary DLBCL of the central nervous system (CNS),or secondary lymphoma of the central nervous system or B-cell lymphomas, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and Burkitt lymphoma, orB-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and classical Hodgkin lymphoma, or primary mediastinal thymic large B-cell lymphomas or primary effusion lymphoma or plasmablastic lymphoma or primary cutaneous DLBCL,leg type or ALK+large B-cell lymphoma or transformed lymphoma or primary testicular DLBCL.
2. Confirmed DLBCL with double (BCL-2 and c-MYC gene rearrangement) or triple (BCL-2, BCL-6, and c-MYC gene rearrangement) hit by FISH. BCL-2 ≥ 70% positive and c-MYC ≥ 40% positive and according to Han's immunohistochemistry method, tumor type is GCB but unable to get unequivocal FISH result.

3．History of other cancers( excluding squamous cell carcinoma of skin, basal cell carcinoma of skin, carcinoma in situ of cervix) within 5 years prior to the enrollment of the study.

4.Patients who received major surgeries (excluding diagnostic surgeries) within 2 months prior to the enrollment of the study.

5. Patients who have received therapy for non-Hodgkin's lymphoma: including chemotherapy, immunotherapy; radiotherapy (excluding local radiotherapy); monoclonal antibody therapy; surgical treatment (excluding biopsy); 6.Patients who received cytotoxic drugs or anti-CD20 monoclonal antibody for other diseases (such as Rheumatoid arthritis).

7. Patients who received any monoclonal antibody within 3 months prior to the enrollment of the study.

8. Patients who participated in other clinical trials within 3 months prior to the enrollment of the study.

9. Patients who received attenuated or live virus vaccine within 1 months prior to the enrollment of the study.

10. Patients who received hematopoietic stimulating factors within 2 weeks prior to the enrollment of the study.

11. Patients who received prednisone>30 mg per day or equivalent corticosteroids for controlling the symptoms other than lymphoma; Patients who received prednisone≤30 mg per day or equivalent corticosteroids should receive stable dose for at least 4 weeks before randomization by written record.

13. Patients with peripheral nervous system or central nervous system disease. 14. Suspected active or latent tuberculosis infections. 15. Within 4 months prior to the enrollment of the study, Patients had active bacteria, virus, fungi, mycobacteria,parasites or other infections(excluding nail bed fungal infection) or in need of intravenous antibiotic treatment or with sever systemic infection or in need of inpatient admission hospital(except for the treatment of neoplastic fever).

16. Other serious diseases that may impair the ability of subjects' participation(e.g., uncontrollable diabetes, (severe cardiac dysfunction, history of myocardial infarction or unstable arrhythmias or unstable angina within the past 6 months or gastric ulcer (gastric ulcer with risk of perforation) or active autoimmune disease or severe hypertension, etc.).

17. Contraindicative to any drug in CHOP, or to anthracycline;Patients with diabetes and intolerant to the prednisone in this study.

18. History of alcohol abuse or drug abuse. 19. Susceptible to allergies or allergic to anyactive ingredients or excipients in the trial (including CHOP) or murine source products ormedication (including CHOP) including active ingredients or excipients or rat source products or heterogeneous proteins.

20. Patients with serious mental disease. 21. Patients who are lack of compliance during the trial and/or the follow-up phase.

22. Patients that researchers deem as not appropriate to enter the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
ORR | 18 weeks
  To evaluate the objective response rate (ORR) in patients with previously untreated Diffuse Large B-cell Lymphoma after six periods of treatment.